CLINICAL TRIAL: NCT04482621
Title: Decitabine for COVID-19 Pneumonia-ARDS Treatment: DART Trial
Brief Title: Decitabine for Coronavirus (COVID-19) Pneumonia- Acute Respiratory Distress Syndrome (ARDS) Treatment: DART Trial
Acronym: DART
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB00247544 is lapsed. Separate application submitted for reactivation under IRB00521868. Awaiting review & approval
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00247544; IRB00521868 (Other: JHM IRB)
Record Dates: First submitted 2020-07-21; First posted 2020-07-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Decitabine

STUDY DESIGN:
Intervention Model Description: This is a randomized double blind placebo controlled Phase 2 trial with a 12 patient lead-in to evaluate safety, prior to full enrollment to an additional 28 patients (for a total of 40 patients) to assess efficacy of decitabine in the treatment of critically ill patients with COVID-ARDS. The patients will be randomized in a 1:1 ratio to receive standard of care plus Decitabine or standard of care plus saline based placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Decitabine + Standard of Care (SOC) (Active Comparator): Study drug Decitabine will be administered via Intravenous injection. Dosage Regimen: 10mg/m^2/day IV day x 5 days (1 cycle only)
  Interventions: Drug: Decitabine
- Standard of Care (SOC) + Placebo (Placebo Comparator): Saline based placebo will be administered via Intravenous injection. Dosage Regimen: 10mg/m^2/day IV day x 5 days (1 cycle only)
  Interventions: Other: Placebo Saline

INTERVENTIONS:
Drug: Decitabine — Study duration is 6 weeks after the last dose of study drug. Number of study visits is dependent on Length of hospitalization of study participant. Study visits are scheduled on days 0-7, 11, 15, 29, and may occur via telemedicine or inpatient assessment or outpatient assessment in COVID recovered participants.
  Decitabine will be administered via Intravenous Administration 10/mg/m^2/day Dosage: 10mg/m^2/day IV day x 5 days (1 cycle only)
  Other Names: 5-aza-2'- deoxycytidine; DACOGEN
  Arms: Decitabine + Standard of Care (SOC)
Other: Placebo Saline — Saline based placebo will be administered via Intravenous injection. Dosage Regimen: 10mg/m^2/day IV day x 5 days (1 cycle only)
  Arms: Standard of Care (SOC) + Placebo

SUMMARY:
This is a a randomized double blind placebo controlled Phase 2 trial with a 12 patient lead-in to evaluate safety, prior to full enrollment to an additional 28 patients (for a total of 40 patients) to assess efficacy of decitabine in the treatment of critically ill patients with COVID-ARDS. The patients will be randomized in a 1:1 ratio to receive standard of care plus Decitabine or standard of care plus saline based placebo. The primary objective is to determine safety and efficacy of decitabine for COVID-19 ARDS based on clinical improvement on a 6-point clinical scale.

DETAILED DESCRIPTION:
This is a randomized double blind placebo controlled Phase 2 trial with a 12 patient lead-in to evaluate safety, prior to full enrollment to an additional 28 patients (for a total of 40 patients) to assess efficacy of decitabine in the treatment of critically ill patients with COVID-ARDS. The patients will be randomized in a 1:1 ratio to receive standard of care plus Decitabine or standard of care plus saline based placebo.

Eligible patients will receive decitabine 10 mg/m2 daily for 5 days, 1 cycle only. This is a dose that is half the FDA approved dose for myelodysplastic syndrome (MDS), and using a single cycle.

If less than 2 of the first 6 (treatment arm) patients experience an unacceptable toxicity, defined as any treatment related grade III or higher adverse events, as per section 5.7, within 15 days of initiation of treatment, the drug is safe to continue. If the investigators observe more than 33% patients with unacceptable toxicity, the investigators will pause the accrual pending safety evaluation. After validating safety, the investigators will enroll additional 28 patients towards the primary efficacy endpoint. The investigators will monitor safety throughout the trial by monitoring clinical hematologic, chemistry, vital signs, respiratory parameters, medications, and clinical changes daily as per the schedule of procedures.

Bio samples from peripheral blood mononuclear cell (PBMC) and Mini Bronchoalveolar lavage (BAL) will be collected and stored for secondary analysis and mini BAL will only be collected as an optional sub-study for patient consented to a separate study protocol either at time-point of for-cause clinically indicated bronchoscopy, or for subjects consented to a separate Bronchoalveolar lavage (BAL) interventional study, under the auspices of that protocol. For research bio specimens required after study drug initiation, a window period of +/-24 hours while inpatient, and +/- 4 days for outpatient monitoring will be permitted.

These objectives will allow for the planning of subsequent phase 3 studies, and strengthen implementation of a multi-center randomized trial should this study confirm safety, and suggest efficacy of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years
2. Use of Intermittent Mechanical Ventilation, non-invasive mechanical ventilation (NIMV) or High Flow Nasal Cannula.
3. Have ARDS or Acute Lung Injury physiology confirmed by Pao2/Fio2 ratio of < 300
4. Severe Acute Respiratory Distress Syndrome (SARS) - Coronavirus (CoV-2) determined by lab polymerase chain reaction assay in either upper or lower respiratory tract sampling (e.g. bronchoalveolar lavage or nasopharyngeal swab)
5. If childbearing age: agree to practice effective birth control from screening until at least 180 days after last dose

Exclusion Criteria:

1. Hematologic cytopenias: Absolute Neutrophil Count (ANC) <1500/mm3, Hgb<7.0 and/or platelets <100,000/mm3
2. Subjects receiving or enrolled in clinical trial for other investigational treatment for SARS- 2-CoV.
3. Active malignancy, solid tumors, and current or recent chemotherapy
4. Concomitant use of nonbiologic immunosuppressants (e.g. Janus Kinase (JAK) inhibitors, Bruton's Tyrosine Kinase (BTK) inhibitors)
5. Active HIV viremia, or any other uncontrolled secondary infection.
6. Concurrent immunomodulating biologics or use of Palifermin, Dipyrone, Deferiprone
7. Subjects with severe sepsis with vasopressors or extrapulmonary organ failure:
8. Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) /alkaline phosphatase (ALK) Phos ≥3x upper limit of normal (ULN) and Total Bilirubin (TBILI) ≥2x ULN; or Creatinine clearance <30 mL/min
9. Pregnant women or women who are breastfeeding
10. Any Condition, per opinion of PI that would affect subject safety and/or compliance
11. Prior hypersensitivity to decitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are alive and free of respiratory failure at day 28 | From the day of randomization to day 28
  The proportion of patients who are alive and free of respiratory failure at day 28 since start of randomization.

SECONDARY OUTCOMES:
Safety as assessed by adverse events | Up to 6 weeks
  Safety assessments using adverse events will be monitored daily while inpatient and weekly through end of study at week 6 once discharged from hospital. They will be monitored and graded using Common Terminology Criteria Adverse Events version 5.0.
Change in oxygenation index | Daily, up to 6 weeks
  Oxygenation index is used to assess severity of hypoxic respiratory failure. (OI = mean airway pressure (MAP) × Fraction of inspired oxygen (FiO2) × 100÷ partial pressure of oxygen (PaO2). This will be measured daily while subject is on mechanical ventilation up to 6 weeks.
Change in fraction of inspired oxygen | Up to day 29
  Fraction of inspired oxygen in the oxygen delivery system during hospital stay. Measured at 8 am daily during hospital stay and then weekly until day 29.
Overall survival | Up to 6 weeks
  Patients status of alive versus death at completion of study follow up period, i.e. 6 weeks from start.
Length of stay in hospital | Till hospital discharge, up to 6 weeks
  Duration of days from baseline to hospital discharge.
Ventilator free days | Up to 6 weeks
  For subjects who received mechanical ventilation, total number of days from baseline to end of study at 6 weeks that subject was not on mechanical or non invasive mechanical ventilation.
Time to Polymerase chain reaction (PCR) negativity | Up to 6 weeks
  If viremic at starting date of decitabine - time from baseline to 1st recorded negative COVID nucleic acid amplification (NAT) based assay, measured in days.
Percentage of patients with National Early Warning Score 2 of 3 or more | Weekly while patient is in hospital, up to 6 weeks
  Determines the degree of illness of a patient and prompts critical care intervention. This composite score includes Respiratory Rate, Temperature, oxygen Saturation, Blood Pressure, Oxygen inspired and cognitive status. This will be measured at baseline and weekly while patient is in hospital.
All-cause mortality at 28 days since randomization | Daily upto day 28
  Total number of death at 28 days since day of randomization
Percentage of change of clinical score based on World Health Organization 9-point scale at day 10 from randomization | Daily from randomization to day 10
  Determine clinical score from randomization date to day 10
Percentage of change of clinical score based on World Health Organization (WHO 9) COVID progression scale | Weekly while patient is in hospital, up to 6 weeks
  Time from randomization to an at least 2-point decrease in clinical score based on WHO 9-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Pali Shah, M.D, Principal Investigator — Johns Hopkins UIniversity
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835
- [Background] Anders NM, Liu J, Wanjiku T, Giovinazzo H, Zhou J, Vaghasia A, Nelson WG, Yegnasubramanian S, Rudek MA. Simultaneous quantitative determination of 5-aza-2'-deoxycytidine genomic incorporation and DNA demethylation by liquid chromatography tandem mass spectrometry as exposure-response measures of nucleoside analog DNA methyltransferase inhibitors. J Chromatogr B Analyt Technol Biomed Life Sci. 2016 Jun 1;1022:38-45. doi: 10.1016/j.jchromb.2016.03.029. Epub 2016 Mar 21. PMID 27082761
- [Background] Qin C, Zhou L, Hu Z, Zhang S, Yang S, Tao Y, Xie C, Ma K, Shang K, Wang W, Tian DS. Dysregulation of Immune Response in Patients With Coronavirus 2019 (COVID-19) in Wuhan, China. Clin Infect Dis. 2020 Jul 28;71(15):762-768. doi: 10.1093/cid/ciaa248. PMID 32161940
- [Background] Wang CH, Liu CY, Wan YL, Chou CL, Huang KH, Lin HC, Lin SM, Lin TY, Chung KF, Kuo HP. Persistence of lung inflammation and lung cytokines with high-resolution CT abnormalities during recovery from SARS. Respir Res. 2005 May 11;6(1):42. doi: 10.1186/1465-9921-6-42. PMID 15888207
- [Background] Park WY, Goodman RB, Steinberg KP, Ruzinski JT, Radella F 2nd, Park DR, Pugin J, Skerrett SJ, Hudson LD, Martin TR. Cytokine balance in the lungs of patients with acute respiratory distress syndrome. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1896-903. doi: 10.1164/ajrccm.164.10.2104013. PMID 11734443
- [Background] Luce JM, Montgomery AB, Marks JD, Turner J, Metz CA, Murray JF. Ineffectiveness of high-dose methylprednisolone in preventing parenchymal lung injury and improving mortality in patients with septic shock. Am Rev Respir Dis. 1988 Jul;138(1):62-8. doi: 10.1164/ajrccm/138.1.62. PMID 3202402
- [Background] Bernard GR, Luce JM, Sprung CL, Rinaldo JE, Tate RM, Sibbald WJ, Kariman K, Higgins S, Bradley R, Metz CA, et al. High-dose corticosteroids in patients with the adult respiratory distress syndrome. N Engl J Med. 1987 Dec 17;317(25):1565-70. doi: 10.1056/NEJM198712173172504. PMID 3317054
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Background] D'Alessio FR, Tsushima K, Aggarwal NR, West EE, Willett MH, Britos MF, Pipeling MR, Brower RG, Tuder RM, McDyer JF, King LS. CD4+CD25+Foxp3+ Tregs resolve experimental lung injury in mice and are present in humans with acute lung injury. J Clin Invest. 2009 Oct;119(10):2898-913. doi: 10.1172/JCI36498. Epub 2009 Sep 21. PMID 19770521
- [Background] Adamzik M, Broll J, Steinmann J, Westendorf AM, Rehfeld I, Kreissig C, Peters J. An increased alveolar CD4 + CD25 + Foxp3 + T-regulatory cell ratio in acute respiratory distress syndrome is associated with increased 30-day mortality. Intensive Care Med. 2013 Oct;39(10):1743-51. doi: 10.1007/s00134-013-3036-3. Epub 2013 Aug 16. PMID 23949701
- [Background] Garibaldi BT, D'Alessio FR, Mock JR, Files DC, Chau E, Eto Y, Drummond MB, Aggarwal NR, Sidhaye V, King LS. Regulatory T cells reduce acute lung injury fibroproliferation by decreasing fibrocyte recruitment. Am J Respir Cell Mol Biol. 2013 Jan;48(1):35-43. doi: 10.1165/rcmb.2012-0198OC. Epub 2012 Sep 20. PMID 23002097
- [Background] Song H, Zhou Y, Li G, Bai J. Regulatory T cells contribute to the recovery of acute lung injury by upregulating Tim-3. Inflammation. 2015;38(3):1267-72. doi: 10.1007/s10753-014-0096-7. PMID 25526715
- [Background] Goodyear OC, Dennis M, Jilani NY, Loke J, Siddique S, Ryan G, Nunnick J, Khanum R, Raghavan M, Cook M, Snowden JA, Griffiths M, Russell N, Yin J, Crawley C, Cook G, Vyas P, Moss P, Malladi R, Craddock CF. Azacitidine augments expansion of regulatory T cells after allogeneic stem cell transplantation in patients with acute myeloid leukemia (AML). Blood. 2012 Apr 5;119(14):3361-9. doi: 10.1182/blood-2011-09-377044. Epub 2012 Jan 10. PMID 22234690
- [Background] Schroeder T, Czibere A, Platzbecker U, Bug G, Uharek L, Luft T, Giagounidis A, Zohren F, Bruns I, Wolschke C, Rieger K, Fenk R, Germing U, Haas R, Kroger N, Kobbe G. Azacitidine and donor lymphocyte infusions as first salvage therapy for relapse of AML or MDS after allogeneic stem cell transplantation. Leukemia. 2013 Jun;27(6):1229-35. doi: 10.1038/leu.2013.7. Epub 2013 Jan 14. PMID 23314834
- [Background] Choi J, Ritchey J, Prior JL, Holt M, Shannon WD, Deych E, Piwnica-Worms DR, DiPersio JF. In vivo administration of hypomethylating agents mitigate graft-versus-host disease without sacrificing graft-versus-leukemia. Blood. 2010 Jul 8;116(1):129-39. doi: 10.1182/blood-2009-12-257253. Epub 2010 Apr 27. PMID 20424188
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Grein J, Ohmagari N, Shin D, Diaz G, Asperges E, Castagna A, Feldt T, Green G, Green ML, Lescure FX, Nicastri E, Oda R, Yo K, Quiros-Roldan E, Studemeister A, Redinski J, Ahmed S, Bernett J, Chelliah D, Chen D, Chihara S, Cohen SH, Cunningham J, D'Arminio Monforte A, Ismail S, Kato H, Lapadula G, L'Her E, Maeno T, Majumder S, Massari M, Mora-Rillo M, Mutoh Y, Nguyen D, Verweij E, Zoufaly A, Osinusi AO, DeZure A, Zhao Y, Zhong L, Chokkalingam A, Elboudwarej E, Telep L, Timbs L, Henne I, Sellers S, Cao H, Tan SK, Winterbourne L, Desai P, Mera R, Gaggar A, Myers RP, Brainard DM, Childs R, Flanigan T. Compassionate Use of Remdesivir for Patients with Severe Covid-19. N Engl J Med. 2020 Jun 11;382(24):2327-2336. doi: 10.1056/NEJMoa2007016. Epub 2020 Apr 10. PMID 32275812
- [Background] Singer BD, Mock JR, Aggarwal NR, Garibaldi BT, Sidhaye VK, Florez MA, Chau E, Gibbs KW, Mandke P, Tripathi A, Yegnasubramanian S, King LS, D'Alessio FR. Regulatory T cell DNA methyltransferase inhibition accelerates resolution of lung inflammation. Am J Respir Cell Mol Biol. 2015 May;52(5):641-52. doi: 10.1165/rcmb.2014-0327OC. PMID 25295995
- [Background] Issa JP, Garcia-Manero G, Giles FJ, Mannari R, Thomas D, Faderl S, Bayar E, Lyons J, Rosenfeld CS, Cortes J, Kantarjian HM. Phase 1 study of low-dose prolonged exposure schedules of the hypomethylating agent 5-aza-2'-deoxycytidine (decitabine) in hematopoietic malignancies. Blood. 2004 Mar 1;103(5):1635-40. doi: 10.1182/blood-2003-03-0687. Epub 2003 Nov 6. PMID 14604977
- [Background] Kantarjian HM, Issa JP. Decitabine dosing schedules. Semin Hematol. 2005 Jul;42(3 Suppl 2):S17-22. doi: 10.1053/j.seminhematol.2005.05.006. PMID 16015500
- [Background] Kantarjian H, Oki Y, Garcia-Manero G, Huang X, O'Brien S, Cortes J, Faderl S, Bueso-Ramos C, Ravandi F, Estrov Z, Ferrajoli A, Wierda W, Shan J, Davis J, Giles F, Saba HI, Issa JP. Results of a randomized study of 3 schedules of low-dose decitabine in higher-risk myelodysplastic syndrome and chronic myelomonocytic leukemia. Blood. 2007 Jan 1;109(1):52-7. doi: 10.1182/blood-2006-05-021162. Epub 2006 Aug 1. PMID 16882708
- [Background] Welch JS, Petti AA, Miller CA, Fronick CC, O'Laughlin M, Fulton RS, Wilson RK, Baty JD, Duncavage EJ, Tandon B, Lee YS, Wartman LD, Uy GL, Ghobadi A, Tomasson MH, Pusic I, Romee R, Fehniger TA, Stockerl-Goldstein KE, Vij R, Oh ST, Abboud CN, Cashen AF, Schroeder MA, Jacoby MA, Heath SE, Luber K, Janke MR, Hantel A, Khan N, Sukhanova MJ, Knoebel RW, Stock W, Graubert TA, Walter MJ, Westervelt P, Link DC, DiPersio JF, Ley TJ. TP53 and Decitabine in Acute Myeloid Leukemia and Myelodysplastic Syndromes. N Engl J Med. 2016 Nov 24;375(21):2023-2036. doi: 10.1056/NEJMoa1605949. PMID 27959731
- [Background] Issa JP, Garcia-Manero G, Huang X, Cortes J, Ravandi F, Jabbour E, Borthakur G, Brandt M, Pierce S, Kantarjian HM. Results of phase 2 randomized study of low-dose decitabine with or without valproic acid in patients with myelodysplastic syndrome and acute myelogenous leukemia. Cancer. 2015 Feb 15;121(4):556-61. doi: 10.1002/cncr.29085. Epub 2014 Oct 21. PMID 25336333
- [Background] Issa JP, Gharibyan V, Cortes J, Jelinek J, Morris G, Verstovsek S, Talpaz M, Garcia-Manero G, Kantarjian HM. Phase II study of low-dose decitabine in patients with chronic myelogenous leukemia resistant to imatinib mesylate. J Clin Oncol. 2005 Jun 10;23(17):3948-56. doi: 10.1200/JCO.2005.11.981. Epub 2005 May 9. PMID 15883410
- [Background] Mock JR, Garibaldi BT, Aggarwal NR, Jenkins J, Limjunyawong N, Singer BD, Chau E, Rabold R, Files DC, Sidhaye V, Mitzner W, Wagner EM, King LS, D'Alessio FR. Foxp3+ regulatory T cells promote lung epithelial proliferation. Mucosal Immunol. 2014 Nov;7(6):1440-51. doi: 10.1038/mi.2014.33. Epub 2014 May 21. PMID 24850425
- [Background] Wijermans P, Lubbert M, Verhoef G, Bosly A, Ravoet C, Andre M, Ferrant A. Low-dose 5-aza-2'-deoxycytidine, a DNA hypomethylating agent, for the treatment of high-risk myelodysplastic syndrome: a multicenter phase II study in elderly patients. J Clin Oncol. 2000 Mar;18(5):956-62. doi: 10.1200/JCO.2000.18.5.956. PMID 10694544
- [Background] Santini V, Kantarjian HM, Issa JP. Changes in DNA methylation in neoplasia: pathophysiology and therapeutic implications. Ann Intern Med. 2001 Apr 3;134(7):573-86. doi: 10.7326/0003-4819-134-7-200104030-00011. PMID 11281740
- [Background] Kaminskas E, Farrell AT, Wang YC, Sridhara R, Pazdur R. FDA drug approval summary: azacitidine (5-azacytidine, Vidaza) for injectable suspension. Oncologist. 2005 Mar;10(3):176-82. doi: 10.1634/theoncologist.10-3-176. PMID 15793220
- [Background] Go L, Budinger GR, Kwasny MJ, Peng J, Forel JM, Papazian L, Jain M. Failure to Improve the Oxygenation Index Is a Useful Predictor of Therapy Failure in Acute Respiratory Distress Syndrome Clinical Trials. Crit Care Med. 2016 Jan;44(1):e40-4. doi: 10.1097/CCM.0000000000001295. PMID 26427588
- [Background] Seeley E, McAuley DF, Eisner M, Miletin M, Matthay MA, Kallet RH. Predictors of mortality in acute lung injury during the era of lung protective ventilation. Thorax. 2008 Nov;63(11):994-8. doi: 10.1136/thx.2007.093658. Epub 2008 Jun 19. PMID 18566110
- [Background] Jabbour E, Short NJ, Montalban-Bravo G, Huang X, Bueso-Ramos C, Qiao W, Yang H, Zhao C, Kadia T, Borthakur G, Pemmaraju N, Sasaki K, Estrov Z, Cortes J, Ravandi F, Alvarado Y, Komrokji R, Sekeres MA, Steensma DP, DeZern A, Roboz G, Kantarjian H, Garcia-Manero G. Randomized phase 2 study of low-dose decitabine vs low-dose azacitidine in lower-risk MDS and MDS/MPN. Blood. 2017 Sep 28;130(13):1514-1522. doi: 10.1182/blood-2017-06-788497. Epub 2017 Aug 3. PMID 28774880
- [Derived] Sinnige JS, Filippini DFL, Hagens LA, Heijnen NFL, Schnabel RM, Schultz MJ, Bergmans DCJJ, Bos LDJ, Smit MR. Associations of early changes in lung ultrasound aeration scores and mortality in invasively ventilated patients: a post hoc analysis. Respir Res. 2024 Jul 8;25(1):268. doi: 10.1186/s12931-024-02893-0. PMID 38978068